CLINICAL TRIAL: NCT04249453
Title: The Assessment of Lower Back Mechanical Behavior and Spinal Loads in Veterans With Non-specific Low Back Pain: a Feasibility Study
Brief Title: Lower Back Biomechanics in Veterans With Non-Specific Low Back Pain
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor
Other Study IDs: F3300-P
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Chronic Low Back Pain
Keywords: Back pain; Lumbar spine; Biomechanics; Spinal loads
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Chronic low back pain with high disability: Veterans with chronic, non-specific LBP and a Roland-Morris Disability Questionnaire (RMDQ) score of >12 (gender-balanced, n1=18)
- Chronic low back pain with low disability: Veterans with chronic, non-specific LBP and a RMDQ score of 12 (gender-balanced, n2=18)
- Controls: Asymptomatic veterans with no recent history of LBP (gender-balanced, n3=18)

SUMMARY:
Low back pain (LBP) is strongly associated with opioid consumption among Veterans, and improved clinical management of LBP is likely to reduce reliance on opioid among Veterans. Up to 60% of patients with an acute episode of nonspecific LBP experience either symptom persistence or symptom relapse within one year. This is likely an indication of a failure in addressing the underlying mechanisms of pain or initiation of a new etiology; both may stem from a mismatch between patients and treatments. The overall goal of this research is to develop, validate and implement measures that are relevant to known mechanisms of LBP, which can then be used to holistically gauge the health status of patients' lower backs beyond self-reporting of symptoms. More accurate measurements will help better match of patients with existing treatments or development of more effective new treatments. The specific objective of this study is to generate evidence in support of the feasibility of the investigators' methods for 1) the evaluation of relative contribution of lower back tissues to spinal loads, and 2) the investigation of the resultant spinal loads in Veterans with non-specific LBP. The investigators have developed a powerful set of tools for the comprehensive assessment of spinal loads and lower back mechanical behavior (MB), that will enable the investigators to examine the existence or development of abnormalities in spinal loads and lower back MB in three groups of Veterans with different experiences with non-specific LBP. These groups will include 1) Veterans with chronic, non-specific LBP and high level of disability (n=18), 2) Veterans with chronic, non-specific LBP and low level of disability (n=18), 3) asymptomatic Veterans without a recent history of non-specific LBP (n=18; serving as control group). Successful completion of this feasibility project will pave the way for future studies (merit grant applications) that will verify the role of abnormalities in lower back MB and spinal loads in the clinical presentation of LBP. Such an understanding has the potential to help the affected Veterans with disabling non-specific LBP. Specifically, measures of lower back MB and spinal loads can be used not only to identify Veterans with mechanical abnormalities in their lower back who are likely to experience LBP in the future, but also to guide novel integrated physical and psychological preventative treatments aimed at improved lower back mechanics. Ultimately, the goal and resultant improvement in clinical outcomes of treatment for non-specific LBP is to diminish reliance on opioids for the symptom management of particularly Veterans with chronic LBP.

DETAILED DESCRIPTION:
Specific Aims

The specific objective of this study is to generate evidence in support of the feasibility of the investigators' developed methods for the evaluation of 1) relative contribution of lower back tissues to spinal loads, and 2) the resultant spinal loads experienced during daily activities in Veterans with non-specific LBP. Results of this feasibility study will enable proper design of the investigators' future projects, wherein the investigators will investigate the role of spinal loads experienced in daily life activities in clinical presentation of LBP. The investigators have developed several innovative computational and experimental methods for a comprehensive and personalized assessment of spinal loads. Specifically, the relative mechanical contribution of active and passive lower back tissues to spinal loads is assessed using advanced measures of bulk lower back mechanical behavior (MB), whereas muscular responses to physical demands of daily activities and the resultant spinal loads are evaluated using the investigators' finite element model of human spine. The investigators have used the methods proposed in this application extensively for evaluation of bulk lower back MB and spinal loads in asymptomatic individuals. This project will demonstrate the sensitivity of the measures for capturing abnormalities in lower back MB and spinal loads in patients with nonspecific LBP by completing the following two aims to achieve the investigators' objective:

Aim-1: Feasibility of distinguishing potential differences in lower back MB between Veterans with different LBP experiences. The investigators will characterize lower back MB in three gender-balanced groups of Veterans between 20 and 70 years old. These will include Veterans with 1) chronic LBP and a Roland-Morris Disability Questionnaire (RMDQ) score of >12 (n=18), 2) chronic LBP and RMDQ score of 12 (n=18), 3) no recent history of LBP and currently asymptomatic (n=18), serving as control group). Participants will be recruited from the population served by the Lexington, KY, VA Medical Center. The investigators will determine passive stiffness of the lower back and its relaxation along with its active intrinsic and reflexive mechanical properties, using the sudden perturbation and stress-relaxations tests. Given the reported differences in trunk neuromuscular behavior and lumbo-pelvic coordination, the investigators expect to see differences in the measures between patient groups targeted for this project.

Aim-2: Feasibility of distinguishing potential differences in spinal loads between Veterans with different LBP experiences. Trunk muscle forces and the resultant spinal loads will be determined in the same participant groups when they perform common activities of daily living like walking and manual material handling. Considering the causal role of spinal loads, and given the persistence of symptom in patients with chronic LBP, along with the high risk of LBP recurrence in patients with non-chronic LBP and those with a recent history of LBP, the investigators expect differences in spinal loads between patient groups.

Research Procedures:

Participants deemed eligible will complete one data collection session during which they will first be instrumented with sensors to enable measurement of kinematics and muscle activity, similar to procedures the investigators used in earlier studies. Specifically, wireless inertial measurement units (Xsens MTW, Xsens Technologies, Enschede, Netherlands) will be used to measure rotations of the thorax and pelvis, and surface EMG electrodes will be used to measure the activity of erector spinae, rectus abdominis, internal and external obliques. Participants will then be asked to stand on a force plate and perform a forward bending and backward return test. Participants will be instructed to bend from an upright standing posture to their maximum comfortable forward bending posture and then return to the upright posture at a self-selected pace. Participants will then be instructed to perform the following activities of daily life at a self-selected pace: walking on level and sloped surfaces, sit-to-stand and stand-to-sit motions, and lowering and lifting a 10 lb load to their knee height. These activities have been selected because they represent basic but repetitive activities of daily life, and the investigators have successfully used them in earlier investigation of spinal loads among asymptomatic non-Veterans, as well as persons with unilateral lower limb amputation. Finally, sudden perturbation followed by stress-relaxation tests will be conducted as in earlier studies and as explained below. Each of the above tests will take less than 5 minutes, and the investigators will provide break periods between each set of tests to minimize fatigue and discomfort.

In preparation for future projects, the investigators will also administer the following questionnaires that are relevant to LBP experience during the data collection session: 1) comprehensive health status using the PROMIS-29 questionnaire (all participants), 2) survey of habitual physical activity (all participants), 3) the short version of Copenhagen Psychosocial questionnaire concerning work and non-work-related factors (all participants), 4) the minimum data set recommended by the NIH task force on research standards for chronic LBP (only Veterans with LBP), 5) pain intensity using a numerical rating scale (only Veterans with LBP), 6) LBP-related disability using the 24-item Roland Morris Disability Questionnaire (only Veterans with LBP), 7) the fear-avoidance beliefs questionnaire (only Veterans with LBP). Total time for the entire data collection session, including the instrumentation time, is estimated to be less than 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 70 years old
* Body mass index between 22 and 32

Exclusion Criteria:

* Any spinal surgery [e.g., spinal fusion surgery]
* Any abnormalities in lower extremity joints due to disease or injury that would likely affects lower back mechanics [e.g., lower limb amputation or peripheral arterial disease]
* Any safety concern [e.g., pregnancy]
* Any medical condition for which we can't determine the impact of the investigators' experimental procedures. [e.g., we don't know whether our measurement instrument will affect pacemakers.]
* Can't complete the tolerability tests for sudden perturbation and stress-relaxation (see description given under "Risk versus benefits")]
* Inability to read or verbally comprehend English
* Unwilling or unable to comply with study protocol
* Retention of legal advice or an open / pending legal case related to LBP

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit 54 gender-balanced veterans in the following three groups: 1) with chronic, non-specific LBP and a Roland-Morris Disability Questionnaire (RMDQ) score of >12 (n=18), 2) with chronic, non-specific LBP and a RMDQ score of =12 (n=18), 3) asymptomatic and no a recent history of non-specific LBP (n=18; serving as control group)
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Estimates of Spinal load from finite element model | Within a week of data collection for each participant, 12-18 month for all participants
  The maximum spinal load experienced at the L5-S1 level during each activity. This measure is estimated by our finite element model. The input to the model will be measurements of trunk and pelvis motion
Reflex delay calculated using measurements of muscle EMG and trunk kinetics | Within a week of data collection for each participant, 12-18 month for all participants
  Latency of reflexive response of trunk muscles to sudden perturbations. This measure will be calculated using a system identification and by relating measured muscle activities (EMG) and trunk kinetics.
Intrinsic stiffness calculated using measurements of trunk kinetics and kinematics | Within a week of data collection for each participant, 12-18 month for all participants
  Intrinsic stiffness refers to aspects of lower back mechanical behavior that are quantified during the reflex delay period (i.e., between perturbation onset and reflexive muscle response), and which incorporate both passive and active contributions of lower back tissues.
Reflexive force calculated using measurements of muscle EMG and trunk kinetics | Within a week of data collection for each participant, 12-18 month for all participants
  The maximum value of reflexive response of trunk muscles to sudden perturbations. To obtain the maximum reflexive force, the reflexive responses of lower back will be estimated by subtracting the intrinsic response from the measured trunk response (i.e., reaction force from load cell) over a time window between the end of latency period and 150 msec post perturbation.
Passive stiffness calculated using measurements of trunk kinetics and kinematics | Within a week of data collection for each participant, 12-18 month for all participants
  Average stiffness of lower back obtained from the stress-relaxation test.
Viscoelastic relaxation calculated using measurements of trunk kinetics and kinematics | Within a week of data collection for each participant, 12-18 month for all participants
  The amount of relaxation in passive resistance of lower back during the stress-relaxation test.

CONTACTS AND LOCATIONS:
Overall Officials: Babak Bazrgari, PhD, Principal Investigator — Lexington VA Medical Center, Lexington, KY
Locations (1):
- Lexington VA Medical Center, Lexington, KY, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT04249453/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT04249453/ICF_001.pdf